CLINICAL TRIAL: NCT02063880
Title: Urgent Versus Post-Stabilization ART in HIV-1 Infected Children With Severe Co-Infections
Brief Title: Pediatric Urgent Start of Highly Active Antiretroviral Treatment (HAART)
Acronym: PUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Nairobi (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001052; 2R01HD023412-21 (NIH)
Record Dates: First submitted 2012-08-21; First posted 2014-02-17 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Human Immunodeficiency Virus; Immune Reconstitution Inflammatory Syndrome
Keywords: HIV-1; IRIS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Immune Reconstitution Inflammatory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Urgent ART (Experimental): Initiation of highly active antiretroviral therapy (HAART) within 48 hours of enrollment.
  Antiretroviral therapy will include regimens recommended by the Kenyan Ministry of Health.
  Interventions: Other: Urgent ART
- Early ART (Active Comparator): Initiation of HAART 7-14 days after enrollment.
  Interventions: Other: Early ART

INTERVENTIONS:
Other: Urgent ART — Children will be started on HAART <48 hours after enrollment.
  Other Names: HAART regimens recommended by WHO and Kenya MOH.
  Arms: Urgent ART
Other: Early ART — Children will be started on ART after stabilization 7-14 days after enrollment.
  Arms: Early ART

SUMMARY:
Design: Randomized clinical trial involving hospitalized HIV-1 infected children. Children will be randomized to randomized to urgent (<48 hours) versus early antiretroviral therapy (7-14 days). This trial will be unblinded.

Population: Hospitalized HIV-1 infected children who are antiretroviral therapy (ART) naïve ≤ 12 years of age.

Sample size: 360 children will be randomized (180 per arm).

Treatment: All infants will be treated with ART according to World Health Organization (WHO) and Kenyan national guidelines.

Study duration: Enrollment into the study will occur over the course of 36-48 months and each infant will be routinely followed for a maximum of 6 months.

Study site: Kenyan hospitals.

Primary hypothesis:

HIV-1 infected children hospitalized with severe co-infection either may be unsalvageable due to too far advanced immunosuppression/co-infection or may benefit from urgent ART.

Secondary hypotheses:

Urgent ART during an acute infection could potentially result in increased risk of immune reconstitution inflammatory syndrome (IRIS) or drug toxicities/interactions.

Specific aims:

1. To compare the 6 month all-cause mortality rate, incidence of immune reconstitution inflammatory syndrome (IRIS), and incidence of drug toxicity in HIV-1 infected children (≤ 12 years old) presenting to hospital with a serious infection randomized to urgent (<48 hours) versus early ART (7-14 days).
2. To determine co-factors for mortality, IRIS, and drug toxicity. Potential cofactors will include: baseline weight-for-age, height-for-age, weight-for-height (Z-scores), CD4, HIV-1 RNA, type of co-infection, age, rate of viral load and CD4 change following ART, immune activation markers, pathogen and HIV-1 specific immune responses.

Secondary aim: To determine etiologies of IRIS and to compare immune reconstitution to HIV, TB, EBV and CMV following ART overall and in each trial arm.

DETAILED DESCRIPTION:
Children will be followed and compared for 6-month mortality.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≤ 12 years old (reported)
* HIV-1 positive (for example, two rapid HIV-1 antibody tests for children >18 months and not breastfeeding, or one HIV-1 DNA/RNA test for children ≤18 months or who are breastfeeding)
* Not currently receiving antiretroviral therapy (history of pMTCT does not affect eligibility)
* Eligible to receive ART, according to current WHO guidelines
* Caregiver plans to reside in study catchment area for at least 6 months (reported)
* Caregiver provides sufficient locator information

Exclusion Criteria:

* Suspected meningitis, any other central nervous system infection, or encephalitis

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace John Stewart, MD, PhD, Principal Investigator — University of Washington
Locations (4):
- Kenya (4):
  - JOOTRH, Kisumu
  - Kisumu District Hospital, Kisumu
  - Mbagathi District Hospital, Nairobi
  - Kenyatta National Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
after primary and secondary outcomes are published

REFERENCES:
- [Derived] Cherkos AS, Cranmer LM, Njuguna I, LaCourse SM, Mugo C, Moraa H, Maleche-Obimbo E, Enquobahrie DA, Richardson BA, Wamalwa D, John-Stewart G. Effect of tuberculosis-HIV co-treatment on clinical and growth outcomes among hospitalized children newly initiating antiretroviral therapy. AIDS. 2024 Mar 15;38(4):579-588. doi: 10.1097/QAD.0000000000003797. Epub 2023 Nov 27. PMID 38016160
- [Derived] Njuguna IN, Cranmer LM, Wagner AD, LaCourse SM, Mugo C, Benki-Nugent S, Richardson BA, Stern J, Maleche-Obimbo E, Wamalwa DC, John-Stewart G. Brief Report: Cofactors of Mortality Among Hospitalized HIV-Infected Children Initiating Antiretroviral Therapy in Kenya. J Acquir Immune Defic Syndr. 2019 Jun 1;81(2):138-144. doi: 10.1097/QAI.0000000000002012. PMID 31095004
- [Derived] LaCourse SM, Cranmer LM, Njuguna IN, Gatimu J, Stern J, Maleche-Obimbo E, Walson JL, Wamalwa D, John-Stewart GC, Pavlinac PB. Urine Tuberculosis Lipoarabinomannan Predicts Mortality in Hospitalized Human Immunodeficiency Virus-Infected Children. Clin Infect Dis. 2018 May 17;66(11):1798-1801. doi: 10.1093/cid/ciy011. PMID 29324985
- [Derived] Njuguna IN, Cranmer LM, Otieno VO, Mugo C, Okinyi HM, Benki-Nugent S, Richardson B, Stern J, Maleche-Obimbo E, Wamalwa DC, John-Stewart GC. Urgent versus post-stabilisation antiretroviral treatment in hospitalised HIV-infected children in Kenya (PUSH): a randomised controlled trial. Lancet HIV. 2018 Jan;5(1):e12-e22. doi: 10.1016/S2352-3018(17)30167-4. Epub 2017 Nov 14. PMID 29150377
- [Derived] Wagner AD, Njuguna IN, Andere RA, Cranmer LM, Okinyi HM, Benki-Nugent S, Chohan BH, Maleche-Obimbo E, Wamalwa DC, John-Stewart GC. Infant/child rapid serology tests fail to reliably assess HIV exposure among sick hospitalized infants. AIDS. 2017 Jul 17;31(11):F1-F7. doi: 10.1097/QAD.0000000000001562. PMID 28609404
- [Derived] Njuguna IN, Wagner AD, Cranmer LM, Otieno VO, Onyango JA, Chebet DJ, Okinyi HM, Benki-Nugent S, Maleche-Obimbo E, Slyker JA, John-Stewart GC, Wamalwa DC. Hospitalized Children Reveal Health Systems Gaps in the Mother-Child HIV Care Cascade in Kenya. AIDS Patient Care STDS. 2016 Mar;30(3):119-24. doi: 10.1089/apc.2015.0239. PMID 27308805

RESULTS

PARTICIPANT FLOW:
Groups:
- Urgent ART: Initiation of highly active antiretroviral therapy (HAART) within 48 hours of enrollment.
  Antiretroviral therapy will include regimens recommended by the Kenyan Ministry of Health.
  Urgent ART: Children will be started on HAART <48 hours after enrollment.
Period: Overall Study
Arm/Group | Urgent ART | Early ART
Started | 90 | 93
Completed | 62 | 66
Not Completed | 28 | 27
Not completed — Death | 21 | 18
Not completed — Lost to Follow-up | 7 | 7
Not completed — Ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Urgent ART | Early ART | Total
Number analyzed (Participants) | 90 | 91 | 181
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 2 [0.9 to 6] | 1.8 [0.8 to 4.5] | 1.9 [0.8 to 4.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 50 | 50 | 100
Region of Enrollment [Number; unit: participants]
  Kenya | 90 | 91 | 181
CD4% [Median (Inter-Quartile Range); unit: %] | 12.5 [9 to 18.3] | 17 [9 to 24] | 14.5 [9 to 22]

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Time Frame: 6 months post-HAART initiation
Measure: Number; unit: participants
Arm/Group | Urgent ART | Early ART
Number analyzed (Participants) | 90 | 91
participants | 21 | 18

2. Secondary Outcome: Number of Participants With Evidence of Immune Reconstitution and Inflammatory Syndrome (IRIS)
Description: Confirmed, possible or likely IRIS based on external independent review
Time Frame: 6 months post-HAART initiation
Measure: Number; unit: participants
Arm/Group | Urgent ART | Early ART
Number analyzed (Participants) | 90 | 91
participants | 10 | 12

3. Secondary Outcome: Number of Participants With Potential Drug Toxicity
Description: Participants with adverse events that are deemed to be potentially related to medications.
Time Frame: 6 months post-HAART initiation
Measure: Number; unit: participants
Arm/Group | Urgent ART | Early ART
Number analyzed (Participants) | 90 | 91
participants | 23 | 15

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Urgent ART | Early ART
All-Cause Mortality (participants affected / at risk) | 21/90 | 18/91
Serious Adverse Events (participants affected / at risk) | 34/90 | 40/91
Other Adverse Events (participants affected / at risk) | 10/90 | 12/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urgent ART (N=90) | Early ART (N=91)
Non-mortality SAE (Infections and infestations) | 13 (13) | 22 (22)
Mortality (Infections and infestations) | 21 (21) | 18 (18)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urgent ART (N=90) | Early ART (N=91)
IRIS (Blood and lymphatic system disorders) | 10 (10) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No